CLINICAL TRIAL: NCT00075205
Title: Clinical Trial of the Cannabinoid CB1 Receptor Antagonist, SR141716 (Rimonabant), to Reduce Voluntary Ethanol Drinking in Healthy, Non-Treatment Seeking Individuals Who Consume Between 20 and 50 Drinks Per Week
Brief Title: Rimonabant to Reduce Alcohol Consumption
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Collaborators: Sanofi-Synthelabo (Industry)
Responsible Party: Regina Clementi
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040072; 04-AA-0072
Record Dates: First submitted 2004-01-05; First posted 2004-01-06 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-06-02

CONDITIONS: Healthy; Alcohol Drinking
Keywords: Alcohol Consumption; Alcohol Treatment; Medication Trial; Craving; Cannabinoids; CB 1 Receptor Antagonist; SR141716; Alcoholism
MeSH Terms: conditions — Alcohol Drinking; Alcoholism | interventions — Rimonabant

INTERVENTIONS:
Drug: SR141716 (Rimonabant)

SUMMARY:
This study will examine whether Rimonabant, a drug that blocks cannabinoid-1 (CB1) receptors in the brain, affects alcohol consumption. Substances called endocannabinoids, which have many of the same effects of marijuana, bind to CB1 receptors. Animal studies show that when CB1 receptors are blocked, the animals consume less alcohol.

Healthy normal volunteers between 21 and 40 years of age who consume between 20 and 40 alcoholic drinks per week, drink at least 4 days a week, and are not seeking treatment for alcoholism may be eligible for this study. Candidates are screened with a medical history, including questions about alcohol and drug use, physical examination, blood and urine tests, breath alcohol test, and electrocardiogram.

Participants are asked about their mental health history and use of alcohol, cigarettes and illicit drugs, and fill out questionnaires evaluating their emotional state and personality. Then, they begin a baseline evaluation in which they call a number at the NIH Clinical Center for 21 days to report how much alcohol they drank that day. One week after starting the baseline evaluation, they are randomly assigned to take either Rimonabant or placebo (a pill with no active ingredient) for 2 weeks. Before starting the drug, they have a urine drug screen and measurement of blood alcohol level. After 1 week on the test medication, they return to the Clinical Center to monitor drug or placebo side effects, if any, and to have a blood alcohol level test, urine drug screen, and blood tests for routine blood chemistries. After 2 weeks on the test medication, they come to the Clinical Center at noon for an alcohol self-administration test. Before the test, they are given a breath alcohol test and a urine drug test. The results of both tests must be negative to continue in the study.

The alcohol self-administration test is videotaped. A heparin lock is placed in a vein in the participant's arm. This small needle remains in the arm for the duration of the study to avoid multiple needle sticks for blood draws. Blood is drawn periodically during the test to determine routine laboratory values, cotinine level (assessment of smoking status), the amount of Rimonabant or placebo in the body, and levels of various hormones. Thirty minutes before the test begins and every 30 minutes during the test, participants complete questionnaires and rating scales regarding their mood and desire to drink. Five minutes before the test be...

DETAILED DESCRIPTION:
Recent studies show that endogenous cannabinoids modulate appetitive behaviors. For example, an antagonist of the CB1 cannabinoid receptor, SR141716, decreases food intake in animals as well as in humans and decreases alcohol consumption in rodent models of voluntary ethanol consumption. In this protocol, individuals consuming between 20 and 40 alcohol drinks per week, and who are not seeking alcohol treatment, will be recruited from the community. Following a one week baseline evaluation, participants will be randomized according to a double-blind design to receive either placebo or SR141716 for two additional weeks prior to being admitted to the hospital to participate in an alcohol self-administration experiment. The design of this experiment has been previously shown by O'Malley et al. (1) to be an effective paradigm to study the effects of medication on alcohol consumption. Following baseline psychological and endocrine measures, participants will receive a priming dose of ethanol designed to raise the breath alcohol levels (BAL) to 0.03 g/dl and then have the opportunity to consume up to eight drinks or to receive $3 dollars for each drink not consumed over a two hour period. It is hypothesized that participants receiving SR141716, compared to those receiving placebo, will have decreased alcohol consumption. Following the study, each participant will be carefully counseled about their alcohol consumption and provided referrals for alcohol treatment.

ELIGIBILITY:
* INCLUSION CRITERIA

Male and female healthy participants, between 21 and 45 years of age.

Weight and Body Mass Index:

Males: between 60 kg and 90 kg; Body Mass Index between 18 and 28.

Females: between 45 kg and 80 kg; Body Mass Index between 18 and 28.

Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).

Normal vital signs after 10 minutes in supine position:

systolic blood pressure between 95 mmHg and 140 mmHg,

diastolic blood pressure between 50 mmHg and 90 mmHg,

heart rate between 45 bpm and 90 bpm.

Normal 12-lead EKG, PR less than 210 ms, QRS less than 120 ms, QTcB(1) less than or equal to 430 ms for male and less than or equal to 450 ms for female (incomplete right bundle branch block can be accepted).

Laboratory results should be within the normal range. Laboratory results which are found to be marginally outside the normal range (i.e., minor variances in the complete blood count (CBC) or electrolytes) will be clinically evaluated for relevance to this protocol. Liver functions must be less than two times normal.

Written informed consent prior to study participation.

Female participants of childbearing capability must use a double contraceptive method (such as oral contraceptives, condom with spermicide or intra-uterine device with spermicide) from the start of the study until two months post medication trial.

Normal dietary habits and willingness to abstain from grapefruit juice consumption during the study. (Grapefruit juice inhibits hepatic enzymes which could potentially interfere with the metabolism of SR141716.)

Must agree to abstain from the use of illicit drugs for the duration of the study.

EXCLUSION CRITERIA:

Any history or presence of significant cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic, hematological, neurologic (including any history of convulsions), systemic, infectious diseases, or psychiatric disorders (i.e., a current diagnosis of major depression, panic disorder, eating disorders, or history of schizophrenia, bipolar disorder, or obsessive compulsive disorder). Individuals who report suicidal ideation or who have a past history of suicide attempts.

Frequent headaches and/or migraine, recurrent nausea and/or vomiting.

Symptomatic hypotension whenever the decrease of blood pressure or asymptomatic postural hypotension defined by a decrease in systolic blood pressure (SBP) equal to or greater than 20 mmHg within two minutes when changing from the supine to the standing position.

Blood donation within three months before administration.

Presence or history of any allergy or unusual reactions to drugs or anesthetics that would suggest the participant could have a problem tolerating SR141716 or placebo.

A participant who, in the judgment of the Investigator, is likely to be non-compliant, is violent when drinking, or is unable to cooperate because of a language problem or poor mental development.

Participant who cannot be contacted in case of emergency.

Currently taking any prescription medications or over-the-counter medications on a regular basis. Participants will be allowed to take an occasional pain medication or an antibiotic, if they get sick during their participation in the protocol.

Excessive consumption of beverages with xanthine bases (greater than 6 cups or glasses/day).

Female participants who have a positive Beta-HCG test (urine and/or plasma) or who are lactating.

Positive reaction to any of the following tests: HBs antigen, anti-HCVantibody, anti-HIV1 antibodies, anti-HIV2 antibodies. (Hepatitis could interfere with the metabolism of SR141716 in the liver. HIV could alter brain function.)

Positive results of screening for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, or opiates).

A DSM-IV diagnosis of illicit drug dependence in the last 6 months.

Participants who come to the NIAAA Clinic and evidence withdrawal symptoms that result in a score of 8 or above on the CIWA Instrument.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2003-12-31; Primary Completion 2007-03-15 (Actual); Study Completion 2007-03-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] O'Malley SS, Krishnan-Sarin S, Farren C, Sinha R, Kreek MJ. Naltrexone decreases craving and alcohol self-administration in alcohol-dependent subjects and activates the hypothalamo-pituitary-adrenocortical axis. Psychopharmacology (Berl). 2002 Feb;160(1):19-29. doi: 10.1007/s002130100919. Epub 2002 Jan 22. PMID 11862370
- [Background] Schwartz MW, Woods SC, Porte D Jr, Seeley RJ, Baskin DG. Central nervous system control of food intake. Nature. 2000 Apr 6;404(6778):661-71. doi: 10.1038/35007534. PMID 10766253
- [Background] Levine AS, Morley JE. Neuropeptide Y: a potent inducer of consummatory behavior in rats. Peptides. 1984 Nov-Dec;5(6):1025-9. doi: 10.1016/0196-9781(84)90165-7. PMID 6549409